CLINICAL TRIAL: NCT00549757
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Determine Whether, in Patients With Type 2 Diabetes at High Risk for Cardiovascular and Renal Events, Aliskiren, on Top of Conventional Treatment, Reduces Cardiovascular and Renal Morbidity and Mortality
Brief Title: Aliskiren Trial in Type 2 Diabetes Using Cardiovascular and Renal Disease Endpoints (Core and Extension Phases)
Acronym: ALTITUDE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of benefit and safety concern
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100E2337; 2007-000860-25 (EudraCT Number)
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease
Keywords: Type 2 diabetes mellitus; renal morbidity and mortality; cardiovascular disease; micro-albuminuria; macro-albuminuria; RAAS; renin inhibitor; Reduced estimated glomerular filtration rate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aliskiren (Experimental): In Core (Double Blind) phase, Aliskiren 150 mg once daily (o.d.) for 4 weeks; then patient was uptitrated to 300 mg o.d. at Visit 5/Week 4 (or 150 mg o.d. if patient could not tolerate target dose of study drug). Visits took place at 1, 4 , 5, 8 and 12 weeks after randomization (Visit 3/Week 0). Subsequent visits were planned every three months until end of core phase.
  With the recommendation of Data Monitoring Committee (DMC), after discontinuation of study drug, a follow up was added as Extension Phase (9 months in average) with no active treatment
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator): In Core (Double Blind) phase, placebo to match aliskiren 150 mg once daily (o.d.) for 4 weeks; from Visit 5/Week 4 placebo to match aliskiren 300 mg o.d. (or placebo to match aliskiren 150 mg if patient could not tolerate target dose of study drug). Visits took place 1, 4 , 5, 8 and 12 weeks after randomization (Visit 3/Week 0). Subsequent visits were planned every three months until end of core phase.
  With the recommendation of Data Monitoring Committee (DMC), after discontinuation of study drug, a follow up was added as Extension Phase (9 months in average) with no active treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg film-coated tablets
  Arms: Aliskiren
Drug: Placebo — Placebo to match aliskiren 150 mg film-coated tablets
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine whether, in patients with type 2 diabetes and pre-existing disease of the heart and the circulatory system and/or the kidney, aliskiren at a target dose of 300 mg once daily (compared to placebo), on top of conventional treatment, reduces death and disease caused by the heart, the circulatory system and the kidney.

AMENDMENT 4 RATIONALE (MARCH 2012) :

Protocol amendment 4 served to address the data monitoring committee recommendation dated 14 Dec 2011 to discontinue study treatment in all participating patients. It also addressed the subsequent Health Authorities request to implement a 12 month safety follow-up period (actual duration was 9 months in average) post study drug discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes and at least one of the following:

  * Macroalbuminuria and an eGFR ≥30 mL/min/1.73 m2
  * Microalbuminuria and a reduced kidney function (eGFR eGFR ≥30 and <60 mL/min/1.73 m2)
  * A history of CV disease (previous MI, previous stroke, heart failure, coronary artery disease, history of percutaneous coronary intervention, angiography proven stenosis ≥50% in at least one coronary artery and a reduced kidney function (eGFR ≥30 and <60 mL/min/1.73 m2)
* Concomitant treatment should follow national guidelines and must include either an Angiotensin-converting-enzyme-inhibitor (ACEi) or an Angiotensin-receptor-blocker (ARB) but not both.

Exclusion Criteria:

* Type 1 diabetes mellitus
* Cardiovascular event or procedure ≤ 3 months prior to Visit 1
* Unstable serum creatinine
* Hypertension: Mean sitting systolic blood pressure (msSBP) ≥ 135 and < 170 mmHg or Mean sitting diastolic blood pressure (msDBP) ≥ 85 and < 110 mmHg unless treated with at least 3 anti-hypertensive medications
* Hypertension msSBP ≥ 170 or msDBP ≥ 110 mmHg
* Baseline Serum Potassium > 5.0 mmol/L
* Patients who are treated with two renin-angiotensin-aldosterone-system-blockers
* Patients with NYHA class III or IV heart failure
* Known renal artery stenosis
* Previous randomization into the AVOID trial (CSPP100C2201)

EXCLUSION SPECIFIC TO THE SAFETY FOLLOW-UP PERIOD:

- Aliskiren or aliskiren containing fixed combination products must not be used

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8606 (Actual)
Dates: Start 2007-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (609):
- United States (102):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Montgomery, Alabama
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Fayetteville, Arkansas
  - Novartis Investigative Site, Burlingame, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Spring Valley, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Bridgeport, Connecticut
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Lauderdale Lakes, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Cumming, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Champaign, Illinois
  - Novartis Investigative Site, Lake Zurich, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Haverhill, Massachusetts
  - Novartis Investigative Site, Jamaica Plain, Massachusetts
  - Novartis Investigative Site, Natick, Massachusetts
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Waltham, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Louis Park, Minnesota
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Gulfport, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Fremont, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Dover, New Hampshire
  - Novartis Investigative Site, Princeton Junction, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Lyndhurst, Ohio
  - Novartis Investigative Site, Norman, Oklahoma
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Allentown, Pennsylvania
  - Novartis Investigative Site, Lancaster, Pennsylvania
  - Novartis Investigative Site, Lansdale, Pennsylvania
  - Novartis Investigative Site, Melrose Park, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Wyomissing, Pennsylvania
  - Novartis Investigative Site, Warwick, Rhode Island
  - Novartis Investigative Site, Aiken, South Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Orangeburg, South Carolina
  - Novartis Investigative Site, Collierville, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Irving, Texas
  - Novartis Investigative Site, McAllen, Texas
  - Novartis Investigative Site, North Richland Hills, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Temple, Texas
  - Novartis Investigative Site, Bennington, Vermont
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Alexandria, Virginia
  - Novartis Investigative Site, Burke, Virginia
  - Novartis Investigative Site, Renton, Washington
  - Novartis Investigative Site, Charleston, West Virginia
  - Novartis Investigative Site, Appleton, Wisconsin
- Argentina (10):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, Zárate, Buenos Aires
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
- Austria (7):
  - Novartis Investigative Site, Vienna, Austria
  - Novartis Investigative Site, Bregenz
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (20):
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, De Pinte
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Ronse
  - Novartis Investigative Site, Seraing
  - Novartis Investigative Site, Sint-Gillis-Waas
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Vilvoorde
  - Novartis Investigative Site, Willebroek
- Brazil (13):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Marília, São Paulo
  - Novartis Investigative Site, Santos, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Canada (29):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Bay Roberts, Newfoundland and Labrador
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Courtice, Ontario
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, North Bay, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Thornhill, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Mirabel, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Pointe-Claire, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
  - Novartis Investigative Site, Ouest-Montreal
- China (24):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Qingdao, Shandong
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Dalian
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (4):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Florida Blanca
  - Novartis Investigative Site, Medellín
- Czechia (10):
  - Novartis Investigative Site, České Budějovice, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Písek
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Prague 4 - Krc
  - Novartis Investigative Site, Prague 5 - Motol
- Denmark (10):
  - Novartis Investigative Site, Copenhagen NV, Denmark
  - Novartis Investigative Site, Roskilde, Denmark
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Frederiksberg
  - Novartis Investigative Site, Gentofte Municipality
  - Novartis Investigative Site, Hillerød
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Slagelse
  - Novartis Investigative Site, Svendborg
- Finland (11):
  - Novartis Investigative Site, Oulu, Finland
  - Novartis Investigative Site, Pori, Finland
  - Novartis Investigative Site, Ekenäs
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Hyvinkää
  - Novartis Investigative Site, Kajaani
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Lohja
  - Novartis Investigative Site, OYS
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Valkeakoski
- France (10):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bondy
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, Lagny-sur-Marne
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
- Germany (42):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Aßlar
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Barsinghausen
  - Novartis Investigative Site, Bensheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Bretten
  - Novartis Investigative Site, Cloppenburg
  - Novartis Investigative Site, Dippoldiswalde
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Fuldatal
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hagen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Ingelheim
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Krefeld
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Messkirch
  - Novartis Investigative Site, Muehldorf Am Inn
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Rehburg-Loccum
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Saint Ingbert - Oberwuerzbach
  - Novartis Investigative Site, Schauenburg-Elgershausen
  - Novartis Investigative Site, Schwabenheim
  - Novartis Investigative Site, Ursensollen
  - Novartis Investigative Site, Wetter
  - Novartis Investigative Site, Wiehl
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Würzburg
- Greece (8):
  - Novartis Investigative Site, Alexandroupoli, Greece
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Thessaloniki, Greece
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Athens - GR
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Pátrai
  - Novartis Investigative Site, Piraeurs
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Hungary (10):
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Zalaegerszeg
- India (16):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh, India
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Banglaore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Bangalore
  - Novartis Investigative Site, Chennai
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Kolkota
  - Novartis Investigative Site, New Delhi
- Italy (44):
  - Novartis Investigative Site, L’Aquila, AQ
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Belluno, BL
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Campobasso, CB
  - Novartis Investigative Site, Caserta, CE
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Cosenza, CS
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Arenzano, GE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Lecco, LC
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Passirana Di Rho, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Casorate Primo, PV
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Stradella, PV
  - Novartis Investigative Site, Ravenna, RA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Cava de' Tirreni, SA
  - Novartis Investigative Site, Mercato San Severino, SA
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Olbia, SS
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Vittorio Veneto, TV
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Venezia, VE
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Isernia
  - Novartis Investigative Site, Napoli
- Japan (27):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Asahi, Chiba
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Toride, Ibaraki
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Aira, Kagoshima-ken
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yatsushiro, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Yao, Osaka
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Ohtsu-city, Shiga
  - Novartis Investigative Site, Shimizu, Shizuoka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
- Lithuania (3):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Netherlands (29):
  - Novartis Investigative Site, Almelo, Netherlands
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Apeldoorn
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Den Helder
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Doetinchem
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Goes
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Hoogeveen
  - Novartis Investigative Site, Hoogwoud
  - Novartis Investigative Site, Losser
  - Novartis Investigative Site, Meppel
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Oude Pekela
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Tiel
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Venlo
  - Novartis Investigative Site, Woerden
  - Novartis Investigative Site, Zwijndrecht
  - Novartis Investigative Site, Zwolle
- Norway (13):
  - Novartis Investigative Site, Fredrikstad, Norway
  - Novartis Investigative Site, Horten, Norway
  - Novartis Investigative Site, Skien, Norway
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Hønefoss
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Spikkestad
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Svelvik
  - Novartis Investigative Site, Tromsø
  - Novartis Investigative Site, Trondheim
  - Novartis Investigative Site, Tønsberg
- Peru (6):
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Santiago de Surco, Lima region
- Portugal (11):
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Lisbon, Portugal
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Linda a Velha
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Portimão
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Santa Maria da Feira
  - Novartis Investigative Site, Santarém
- Novartis Investigative Site, Ponce, Puerto Rico
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- Slovakia (14):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Žilina, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Nitra, Slovakia
  - Novartis Investigative Site, Banksa Bystrica
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Ľubochňa
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Prievidza
  - Novartis Investigative Site, Trstená
- South Africa (7):
  - Novartis Investigative Site, Somerset West, Western Cape
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Gauteng
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Port Elizabeth
  - Novartis Investigative Site, Pretoria
- South Korea (10):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Ansan, Gyeonggi-do
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Bundang, Seongnam
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (52):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, El Puerto de Santa María, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Jerez de la Frontera, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Plentzia, Basque Country
  - Novartis Investigative Site, Villabona, Basque Country
  - Novartis Investigative Site, Zumarraga, Basque Country
  - Novartis Investigative Site, Aranda de Duero, Castille and León
  - Novartis Investigative Site, Miranda de Ebro, Castille and León
  - Novartis Investigative Site, Alcázar de San Juan, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, La Pobla Llarga, Catalonia
  - Novartis Investigative Site, Llança, Catalonia
  - Novartis Investigative Site, Manresa, Catalonia
  - Novartis Investigative Site, Mollet del Vallès, Catalonia
  - Novartis Investigative Site, Rubí, Catalonia
  - Novartis Investigative Site, Santa Coloma de Gramanet, Catalonia
  - Novartis Investigative Site, Tàrrega, Catalonia
  - Novartis Investigative Site, Vic, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Begonte, Galicia
  - Novartis Investigative Site, Ferrol, Galicia
  - Novartis Investigative Site, Pontevedra, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Galicia
  - Novartis Investigative Site, Alfaro, La Rioja
  - Novartis Investigative Site, Logroño, La Rioja
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Arganda, Madrid
  - Novartis Investigative Site, Civdad Real, Madrid
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Murcia, Madrid
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Alaquàs, Valencia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Benidorm, Valencia
  - Novartis Investigative Site, Port de Sagunt, Valencia
  - Novartis Investigative Site, Quart de Poblet, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Xixona, Valencia
  - Novartis Investigative Site, Hospitalet de Llbregat
  - Novartis Investigative Site, L'Hospitalet de Llobregat
- Sweden (8):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Helsingborg
  - Novartis Investigative Site, Karlstad
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Rättvik
  - Novartis Investigative Site, Stenstorp
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Varberg
- Switzerland (14):
  - Novartis Investigative Site, Estavayer-le-Lac, CH
  - Novartis Investigative Site, Bolligen, Switzerland
  - Novartis Investigative Site, Winterthur, Switzerland
  - Novartis Investigative Site, Ascona
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Bruderholz
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, La Chaux-de-Fonds
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Renens
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Schaffhausen
  - Novartis Investigative Site, Zurich
- Taiwan (9):
  - Novartis Investigative Site, Yungkang, Tainan
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Niaosong Township
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taichung County
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Altunizade
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
- United Kingdom (20):
  - Novartis Investigative Site, High Wycombe, Buckinghamshire
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Paignton, Devon
  - Novartis Investigative Site, Cornwall, England
  - Novartis Investigative Site, Welwyn Garden City, Hertfordshire
  - Novartis Investigative Site, Gravesend, Kent
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, East Horsley, Surrey
  - Novartis Investigative Site, Crawley, West Sussex
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Irvine
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Merseyside
  - Novartis Investigative Site, Rugby
  - Novartis Investigative Site, Vale of Glanmorgan
  - Novartis Investigative Site, Wrexham
- Venezuela (4):
  - Novartis Investigative Site, Puerto Ordaz and San Felix, Bolívar
  - Novartis Investigative Site, Valencia, Carabobo
  - Novartis Investigative Site, Caracas, Distrito Federal
  - Novartis Investigative Site, Caracas, Miranda

REFERENCES:
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Malachias MVB, Jhund PS, Claggett BL, Wijkman MO, Bentley-Lewis R, Chaturvedi N, Desai AS, Haffner SM, Parving HH, Prescott MF, Solomon SD, De Zeeuw D, McMurray JJV, Pfeffer MA. NT-proBNP by Itself Predicts Death and Cardiovascular Events in High-Risk Patients With Type 2 Diabetes Mellitus. J Am Heart Assoc. 2020 Oct 20;9(19):e017462. doi: 10.1161/JAHA.120.017462. Epub 2020 Sep 23. PMID 32964800
- [Derived] Heerspink HJ, Persson F, Brenner BM, Chaturvedi N, Brunel P, McMurray JJ, Desai AS, Solomon SD, Pfeffer MA, Parving HH, de Zeeuw D. Renal outcomes with aliskiren in patients with type 2 diabetes: a prespecified secondary analysis of the ALTITUDE randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Apr;4(4):309-17. doi: 10.1016/S2213-8587(15)00469-6. Epub 2016 Jan 14. PMID 26774608
- [Derived] Parving HH, Brenner BM, McMurray JJ, de Zeeuw D, Haffner SM, Solomon SD, Chaturvedi N, Persson F, Desai AS, Nicolaides M, Richard A, Xiang Z, Brunel P, Pfeffer MA; ALTITUDE Investigators. Cardiorenal end points in a trial of aliskiren for type 2 diabetes. N Engl J Med. 2012 Dec 6;367(23):2204-13. doi: 10.1056/NEJMoa1208799. Epub 2012 Nov 3. PMID 23121378
- [Derived] Lambers Heerspink HJ, Perkovic V, de Zeeuw D. Renal and cardio-protective effects of direct renin inhibition: a systematic literature review. J Hypertens. 2009 Dec;27(12):2321-31. doi: 10.1097/HJH.0b013e3283310f92. PMID 19727007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per data monitoring committee (DMC) recommendation all patients were required to permanently stop study medication by 06Jan2012. A follow-up period (actual duration, 9 months in average) post study drug discontinuation on 7590 patients was implemented upon request of Health Authority following the recommendation of DMC to cease study treatment.
Period: Active Treatment Phase: Max. 50 Months
Arm/Group | Aliskiren | Placebo
Started | 4296 ("Started" indicates randomized patients.) | 4310
Full Analysis Set | 4274 | 4287
Safety Set | 4272 | 4285
Completed | 0 | 0
Not Completed | 4296 | 4310
Not completed — Adverse Event | 590 | 462
Not completed — Abnormal laboratory value(s) | 98 | 58
Not completed — Abnormal test procedure result(s) | 7 | 7
Not completed — Unsatisfactory therapeutic effect | 47 | 53
Not completed — Subject withdrew consent | 38 | 38
Not completed — Lost to Follow-up | 41 | 29
Not completed — Administrative problems | 2857 | 3019
Not completed — Death | 188 | 200
Not completed — Patient's request | 353 | 380
Not completed — Incorrect Entry | 69 | 55
Not completed — Missing data | 8 | 9
Period: Extension Period (in Average 9 Months)
Arm/Group | Aliskiren | Placebo
Started | 3773 (As explained in "pre-assignment detail", follow up was made after drug discontinuation) | 3817 (As explained in "pre-assignment detail", follow up was made after drug discontinuation)
Completed | 3148 | 3182
Not Completed | 625 | 635
Not completed — Death | 143 | 136
Not completed — Lost to Follow-up | 52 | 47
Not completed — Withdrawal by Subject | 9 | 16
Not completed — Patient's request | 421 | 436

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) : All patients randomized except mis-randomized patients who did not receive study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 4274 | 4287 | 8561
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (9.62) | 64.4 (9.87) | 64.5 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1393 | 1342 | 2735
  Male | 2881 | 2945 | 5826

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Occurrence of Primary Composite Endpoint (Core : Active Treatment Phase)
Description: Occurrence was defined as the first event of the following composite primary endpoint:
  * Cardiovascular (CV) death
  * Resuscitated sudden death
  * Non-fatal myocardial infarction (MI)
  * Non-fatal stroke
  * Unplanned hospitalization for heart failure (HF)
  * Onset of end-stage renal disease (ESRD) or death due to renal failure. Onset of ESRD was defined as initiation of dialysis, renal transplantation, or a serum creatinine concentration above 6.0 mg/dL (530 μmol/L), sustained for at least a month.
  * Doubling of baseline serum creatinine concentration, sustained for at least one month. To fulfill the endpoint, the serum creatinine concentration had to be above the upper limit of normal for men and women according to the central laboratory. The upper limit of normal for men is 1.20 mg/dL and for women is 0.91 mg/dL.
Time Frame: Time from randomization to the first event (Maximum 50 months)
Population: Full Analysis Set (FAS) - All patients randomized except mis-randomized patients who did not receive study drug. Mis-randomized patients were defined as not qualified for randomization and were inadvertently randomized into the study.
Measure: Number; unit: percentage of participants
Groups:
- Aliskiren: In Core (Double Blind) phase, Aliskiren 150 mg once daily (o.d.) for 4 weeks; then patient was uptitrated to 300 mg o.d. at Visit 5/Week 4 (or 150 mg o.d. if patient could not tolerate target dose of study drug). Visits took place at 1, 4 , 5, 8 and 12 weeks after randomization (Visit 3/Week 0). Subsequent visits were planned every three months until end of core phase.
- Placebo: In Core (Double Blind) phase, placebo to match aliskiren 150 mg once daily (o.d.) for 4 weeks; from Visit 5/Week 4 placebo to match aliskiren 300 mg o.d. (or placebo to match aliskiren 150 mg if patient could not tolerate target dose of study drug). Visits took place 1, 4 , 5, 8 and 12 weeks after randomization (Visit 3/Week 0). Subsequent visits were planned every three months until end of core phase.
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 17.6 | 16.3

2. Primary Outcome: Percentage of Participants With Cardiovascular (CV) Death (Core: Active Treatment Phase)
Time Frame: Time from randomization to the first event (Maximum 50 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 5.5 | 4.8

3. Primary Outcome: Percentage of Participants With Resuscitated Sudden Death (Core: Active Treatment Phase)
Description: Resuscitated sudden death was adjudicated when a subject experiences sudden death or cardiac arrest and is successfully resuscitated by cardioversion, defibrillation or cardiopulmonary resuscitation with a meaningful recovery of consciousness. This definition excludes known transient losses of consciousness such as seizure or vasovagal episodes that do not reflect significant cardiac dysfunction.
Time Frame: Time from randomization to the first event (Maximum 50 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 0.4 | 0.2

4. Primary Outcome: Percentage of Participants With Fatal/Non-fatal Myocardial Infarction (MI) (Core: Active Treatment Phase)
Time Frame: Time from randomization to the first event (Maximum 50 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 3.3 | 3.2

5. Primary Outcome: Percentage of Participants With Fatal/Non-fatal Stroke (Core: Active Treatment Phase)
Time Frame: Time from randomization to the first event (Maximum 50 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 3.4 | 2.7

6. Primary Outcome: Percentage of Participants With Onset of End-stage Renal Disease (ESRD) (Core: Active Treatment Phase)
Description: ESRD is defined as initiation of dialysis, renal transplantation, or a serum creatinine concentration above 6.0 mg/dL (530 µmol per liter) or renal death
Time Frame: Time from randomization to the first event (Maximum 50 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 2.7 | 2.5

7. Secondary Outcome: Percentage of Participants With Occurrence of Secondary Cardiovascular Composite Endpoint (Core: Active Treatment Phase)
Description: Occurrence was defined as the first event of the following secondary cardiovascular composite endpoint:
  * Cardiovascular (CV) death
  * Resuscitated sudden death
  * Non-fatal myocardial infarction (MI)
  * Non-fatal stroke
  * Unplanned hospitalization for heart failure (HF)
Time Frame: Time from randomization to the first event (Maximum 50 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 13.4 | 12.1

8. Secondary Outcome: Percentage of Participants With Occurrence of Secondary Renal Composite Endpoint (Core: Active Treatment Phase)
Description: Occurrence was defined as the first event of the following secondary renal composite endpoint:
  * Onset of end-stage renal disease (ESRD) or death due to renal failure. Onset of ESRD was defined as initiation of dialysis, renal transplantation, or a serum creatinine concentration above 6.0 mg/dL (530 μmol/L), sustained for at least a month.
  * Doubling of baseline serum creatinine concentration, sustained for at least one month. To fulfill the endpoint, the serum creatinine concentration had to be above the upper limit of normal for men and women according to the central laboratory.The upper limit of normal for men is 1.20 mg/dL and for women is 0.91 mg/dL.
Time Frame: Time from randomization to the first event (Maximum 50 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 5.6 | 5.5

9. Secondary Outcome: Percentage of Participants With Occurrence of Secondary Cardiovascular Composite Endpoint (Extension Phase)
Description: as for outcome 7
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: Extension-phase Analysis Set (EAS) - All patients who had at least one scheduled or unscheduled visit or who died post cut-off date 20-Dec-2011/end of treatment (EOT).
Measure: Number; unit: percentage of participants
Groups:
- Aliskiren; Placebo: With the recommendation of Data Monitoring Committee (DMC), after discontinuation of study drug, a follow up was added as Extension Phase (9 months in average) with no active treatment.
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 5.0 | 4.8

10. Secondary Outcome: Percentage of Participants With Occurrence of Secondary Renal Composite Endpoint (Extension Phase)
Description: Occurrence was defined as the first event of the following secondary renal composite endpoint:
  * Onset of end-stage renal disease (ESRD) or death due to renal failure. Onset of ESRD was defined as initiation of dialysis, renal transplantation, or a serum creatinine concentration above 6.0 mg/dL (530 μmol/L), sustained for at least a month.
  * Doubling of baseline serum creatinine concentration, sustained for at least one month. To fulfill the endpoint, the serum creatinine concentration had to be above the upper limit of normal for men and women according to the central laboratory. The upper limit of normal for men is 1.20 mg/dL and for women is 0.91 mg/dL.
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 3.3 | 3.6

11. Primary Outcome: Percentage of Participants With Doubling of Baseline Serum Creatinine Concentration, Sustained for at Least One Month (Core: Active Treatment Phase)
Description: To fulfill the endpoint, the serum creatinine concentration had to be above the upper limit of normal for men and women according to the central laboratory. The upper limit of normal for men is 1.20 mg/dL and for women is 0.91 mg/dL.
Time Frame: Time from randomization to the first event (Maximum 50 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 4.6 | 4.7

12. Primary Outcome: Percentage of Participants With Unplanned Hospitalization for Heart Failure (Core: Active Treatment Phase)
Time Frame: Time from randomization to the first event (Maximum 50 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 4.7 | 5.0

13. Primary Outcome: Percentage of Participants With All Cause Mortality (Core: Active Treatment Phase)
Time Frame: Time from randomization to the first event (Maximum 50 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
percentage of participants | 8.4 | 8.0

14. Primary Outcome: Percentage of Participants With Occurrence of Primary Composite Endpoint (Extension Phase)
Description: as for outcome 1
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: Extension-phase Analysis Set (EAS) - All patients who had at least one scheduled or unscheduled visit or who died post cut-off date 20-Dec-2011/EOT.
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 8.0 | 8.0

15. Primary Outcome: Percentage of Participants With Cardiovascular (CV) Death (Extension Phase)
Time Frame: from cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 2.1 | 1.9

16. Primary Outcome: Percentage of Participants With Resuscitated Sudden Death (Extension Phase)
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 0.1 | 0.1

17. Primary Outcome: Percentage of Participants Fatal/Non-fatal Myocardial Infarction (MI) (Extension Phase)
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 month in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 1.4 | 1.1

18. Primary Outcome: Percentage of Participants With Fatal/Non-fatal Stroke (Extension Phase)
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 0.9 | 1.0

19. Primary Outcome: Percentage of Participants With Onset of End-stage Renal Disease (ESRD) (Extension Phase)
Description: as for outcome 6
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 1.4 | 1.5

20. Primary Outcome: Percentage of Participants Doubling of Baseline Serum Creatinine Concentration, Sustained for at Least One Month (Extension Phase)
Description: as for outcome 11
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 2.4 | 2.5

21. Primary Outcome: Percentage of Participants With Unplanned Hospitalization for Heart Failure (Extension Phase)
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 1.7 | 1.5

22. Primary Outcome: Percentage of Participants With All Cause Mortality (Extension Phase)
Time Frame: from cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants | 3.8 | 3.6

23. Other Pre Specified Outcome: Percentage of Participants With Angioedema/Angioedema-like or Colorectal Events (Core : Active Treatment Phase)
Description: AEs of special interest were reported according to a post-marketing commitment to Health Authorities and included angioedema/angioedema-like events and colorectal events/ procedures
Time Frame: Time from randomization to the first event (Maximum 50 months)
Population: Safety Set (SAF) - All patients who received at least one dose of trial medication. Patients were analyzed according to the treatment they received.
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4272 | 4285
percentage of participants
  Angioedema / angioedema-like events | 4.4 | 4.8
  Colorectal events | 2.4 | 2.4

24. Other Pre Specified Outcome: Change From Baseline in Urinary Albumin to Creatinine Ratio (UACR) to Month 6 and to Last Measurement (Core : Active Treatment Phase)
Description: Baseline is the geometric mean of last 3 measurements before visit 3, Post-baseline value is the geometric mean of last 3 measurements during each visit.
  Change from Baseline = Post - Baseline.
Time Frame: Baseline, Month 6 , last measurement (maximum at 50 months)
Population: Full Analysis Set (FAS) - All patients randomized except mis-randomized patients who did not receive study drug. Last observation carried forward (LOCF) computation technique was used for month 6 data. At each visit, only patients with values at both baseline and this time point are included.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/mmol
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4274 | 4287
mg/mmol
  Baseline to Month 6 (n= 4021, 4040) | 0.841 [0.820 to 0.862] | 0.945 [0.922 to 0.968]
  Baseline to Last Measurement (n= 4045, 4080) | 0.872 [0.842 to 0.903] | 1.043 [1.009 to 1.079]

25. Other Pre Specified Outcome: Mean Changes in Estimated Glomerular Filtration Rate (eGFR) From Baseline to Month 3 and Month 6 (Core : Active Treatment Phase)
Description: The eGFR calculation was based on the Abbreviated Modification of Diet in Renal Disease (MDRD) Study Equation. Using this method, the applicable MDRD formula to calculate eGFR was as follows:
  Estimated GFR (mL/min/1.73 m^2) = 175 x (serum creatinine in mg/dL) -1.154 x (Age in years) -0.203 x (0.742 if female) x (1.210 if Black)
  Mean changes in eGFR from baseline to month 3 and month 6 were included for analysis. The LS Mean and Standard Error were based on an ANCOVA repeated-measure model with treatment, visit, treatment-by-visit and baseline eGFR as effect terms.
Time Frame: Baseline to Month 3 and Month 6
Population: Full Analysis Set (FAS) - All patients randomized except mis-randomized patients who did not receive study drug. At each visit (baseline, Month 3 and Month 6) , only patients with values at both baseline and post-baseline time point are included.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 4113 | 4130
mL/min/1.73 m^2 | -2.048 (0.15) | -0.825 (0.15)

26. Other Pre Specified Outcome: Percentage of Participants With Angioedema/Angioedema-like Events or Colorectal Events (Extension Phase)
Description: as for outcome 23
Time Frame: From cut-off date (20Dec2011/End of Treatment (EOT) ) to the first event after cut-off date (9 months in average)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 3773 | 3817
percentage of participants
  Angioedema/ Angioedema-like event | 0.8 | 1.2
  Colorectal events | 0.7 | 0.8

ADVERSE EVENTS:
Groups:
- Core-phase: Aliskiren: In Core (Double Blind) phase, Aliskiren 150 mg once daily (o.d.) for 4 weeks; then patient was uptitrated to 300 mg o.d. at Visit 5/Week 4 (or 150 mg o.d. if patient could not tolerate target dose of study drug). Visits took place at 1, 4 , 5, 8 and 12 weeks after randomization (Visit 3/Week 0). Subsequent visits were planned every three months until end of core phase.
- Core-phase: Placebo: In Core (Double Blind) Phase, Placebo to match aliskiren 150 mg once daily (o.d.) for 4 weeks; from Visit 5/Week 4 placebo to match aliskiren 300 mg o.d. (or placebo to match aliskiren 150 mg if patient could not tolerate target dose of study drug). Visits took place 1, 4 , 5, 8 and 12 weeks after randomization (Visit 3/Week 0). Subsequent visits were planned every three months until final closure of the study.
- Extension-phase: Aliskiren; Extension-phase: Placebo: With the recommendation of Data Monitoring Committee (DMC), after discontinuation of study drug, a follow up was added as Extension Phase (9 months in average) with no active treatment.
Arm/Group | Core-phase: Aliskiren | Core-phase: Placebo | Extension-phase: Aliskiren | Extension-phase: Placebo
Serious Adverse Events (participants affected / at risk) | 1988/4272 | 1893/4285 | 704/3773 | 682/3817
Other Adverse Events (participants affected / at risk) | 3205/4272 | 3069/4285 | 995/3773 | 1023/3817
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core-phase: Aliskiren (N=4272) | Core-phase: Placebo (N=4285) | Extension-phase: Aliskiren (N=3773) | Extension-phase: Placebo (N=3817)
Anaemia (Blood and lymphatic system disorders) | 55 | 36 | 13 | 16
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 7 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 27 | 34 | 5 | 7
Acute left ventricular failure (Cardiac disorders) | 4 | 3 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 48 | 64 | 21 | 19
Angina pectoris (Cardiac disorders) | 93 | 85 | 22 | 22
Angina unstable (Cardiac disorders) | 52 | 43 | 10 | 11
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 5 | 5 | 1 | 0
Arrhythmia (Cardiac disorders) | 10 | 13 | 1 | 3
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 10 | 9 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 59 | 64 | 6 | 17
Atrial flutter (Cardiac disorders) | 12 | 6 | 6 | 1
Atrial tachycardia (Cardiac disorders) | 2 | 1 | 1 | 0
Atrioventricular block (Cardiac disorders) | 5 | 5 | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 15 | 10 | 4 | 2
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 6 | 6 | 2 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 16 | 15 | 2 | 4
Bundle branch block left (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac amyloidosis (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 30 | 23 | 7 | 5
Cardiac asthma (Cardiac disorders) | 2 | 2 | 2 | 1
Cardiac disorder (Cardiac disorders) | 2 | 1 | 2 | 0
Cardiac failure (Cardiac disorders) | 173 | 173 | 67 | 50
Cardiac failure acute (Cardiac disorders) | 14 | 16 | 4 | 3
Cardiac failure chronic (Cardiac disorders) | 14 | 15 | 2 | 6
Cardiac failure congestive (Cardiac disorders) | 90 | 71 | 18 | 21
Cardiac fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 1 | 2 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 12 | 13 | 2 | 3
Cardiogenic shock (Cardiac disorders) | 6 | 8 | 1 | 4
Cardiomegaly (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 2 | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 2 | 4 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1 | 2 | 1
Coronary artery disease (Cardiac disorders) | 67 | 71 | 25 | 20
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 7 | 4 | 0 | 3
Coronary artery stenosis (Cardiac disorders) | 13 | 13 | 3 | 2
Diastolic dysfunction (Cardiac disorders) | 3 | 2 | 0 | 0
Dilatation ventricular (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 2 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 5 | 1 | 2 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 7 | 4 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 5 | 3 | 3 | 0
Left ventricular failure (Cardiac disorders) | 8 | 10 | 3 | 2
Left ventricular hypertrophy (Cardiac disorders) | 2 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 4 | 1 | 1 | 2
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 87 | 65 | 23 | 30
Myocardial ischaemia (Cardiac disorders) | 37 | 35 | 8 | 8
Nodal arrhythmia (Cardiac disorders) | 1 | 2 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 4 | 5 | 0 | 1
Pericardial effusion (Cardiac disorders) | 5 | 6 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0 | 0 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 2 | 2 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 8 | 5 | 4 | 4
Silent myocardial infarction (Cardiac disorders) | 1 | 3 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 4 | 3 | 1 | 0
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 1 | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 5 | 6 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Trifascicular block (Cardiac disorders) | 1 | 1 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 3 | 0 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 3 | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 10 | 5 | 1 | 3
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 7 | 3 | 0 | 4
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0
Congenital arterial malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Familial hypocalciuric hypercalcaemia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Haemoglobinopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 2 | 2 | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 2 | 0 | 0
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 2 | 2 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 3 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 17 | 9 | 1 | 4
Vertigo positional (Ear and labyrinth disorders) | 2 | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 2 | 1 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 1
Cushing's syndrome (Endocrine disorders) | 1 | 0 | 0 | 1
Goitre (Endocrine disorders) | 4 | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 4 | 0 | 0
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0
Primary hyperaldosteronism (Endocrine disorders) | 0 | 1 | 0 | 0
Amaurosis (Eye disorders) | 0 | 1 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 33 | 32 | 12 | 6
Cataract diabetic (Eye disorders) | 1 | 0 | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 1 | 0
Cataract subcapsular (Eye disorders) | 0 | 0 | 0 | 1
Corneal degeneration (Eye disorders) | 0 | 2 | 0 | 0
Cystoid macular oedema (Eye disorders) | 1 | 0 | 0 | 0
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 | 1 | 0 | 0
Diabetic eye disease (Eye disorders) | 1 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 23 | 18 | 2 | 4
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Ectropion (Eye disorders) | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 3 | 1 | 2 | 0
Eyelid oedema (Eye disorders) | 2 | 2 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 4 | 2 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 0 | 0
Iris adhesions (Eye disorders) | 0 | 1 | 0 | 0
Lenticular opacities (Eye disorders) | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 1
Macular fibrosis (Eye disorders) | 4 | 3 | 1 | 0
Macular hole (Eye disorders) | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 0 | 2 | 0 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0 | 0
Optic neuropathy (Eye disorders) | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 2 | 2 | 0 | 0
Pterygium (Eye disorders) | 1 | 0 | 0 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 6 | 6 | 0 | 0
Retinal haemorrhage (Eye disorders) | 4 | 5 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 2 | 0 | 0
Retinopathy (Eye disorders) | 3 | 4 | 0 | 1
Retinopathy proliferative (Eye disorders) | 1 | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Vitreous adhesions (Eye disorders) | 0 | 1 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 17 | 11 | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 13 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 2 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 4 | 2 | 0
Colitis (Gastrointestinal disorders) | 4 | 5 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 4 | 7 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diabetic enteropathy (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diabetic gastroenteropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 15 | 4 | 4
Diverticular perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Duodenal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 5 | 5 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 | 5 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 4 | 3 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Gastric mucosa erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 7 | 12 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 10 | 16 | 2 | 3
Gastritis atrophic (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 2 | 3 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 | 14 | 5 | 3
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4 | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 4 | 3 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 3 | 2 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 5 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 3 | 3 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 8 | 9 | 2 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal angina (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 4 | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ischaemic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 17 | 17 | 2 | 6
Lip oedema (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 5 | 5 | 3 | 0
Mesenteric occlusion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 11 | 8 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 5 | 4 | 4 | 1
Pancreatitis acute (Gastrointestinal disorders) | 8 | 5 | 1 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 8 | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Sciatic hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Stress ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 11 | 0 | 2
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Volvulus (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 22 | 18 | 0 | 2
Adverse drug reaction (General disorders) | 0 | 1 | 1 | 0
Asthenia (General disorders) | 15 | 4 | 6 | 5
Cardiac death (General disorders) | 8 | 7 | 3 | 2
Catheter site haemorrhage (General disorders) | 0 | 0 | 2 | 0
Chest discomfort (General disorders) | 2 | 1 | 0 | 0
Chest pain (General disorders) | 4 | 7 | 4 | 1
Chills (General disorders) | 2 | 0 | 0 | 0
Death (General disorders) | 21 | 15 | 13 | 17
Device battery issue (General disorders) | 0 | 1 | 0 | 1
Device dislocation (General disorders) | 1 | 0 | 0 | 0
Device electrical finding (General disorders) | 1 | 0 | 1 | 0
Device failure (General disorders) | 1 | 0 | 1 | 0
Device lead issue (General disorders) | 1 | 0 | 0 | 1
Device malfunction (General disorders) | 3 | 1 | 1 | 1
Discomfort (General disorders) | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Drug intolerance (General disorders) | 1 | 1 | 0 | 0
Face oedema (General disorders) | 11 | 10 | 2 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0
Fat tissue increased (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 3 | 1 | 0
General physical health deterioration (General disorders) | 2 | 4 | 2 | 2
General symptom (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 10 | 11 | 5 | 3
Granuloma (General disorders) | 1 | 0 | 0 | 0
Hyperplasia (General disorders) | 0 | 1 | 0 | 0
Hyperthermia (General disorders) | 1 | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 1 | 0 | 1
Inflammation (General disorders) | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 0
Localised oedema (General disorders) | 2 | 3 | 2 | 0
Malaise (General disorders) | 2 | 4 | 1 | 0
Medical device complication (General disorders) | 1 | 1 | 1 | 0
Multi-organ failure (General disorders) | 0 | 5 | 4 | 3
Non-cardiac chest pain (General disorders) | 37 | 39 | 8 | 2
Oedema (General disorders) | 2 | 1 | 0 | 0
Oedema due to cardiac disease (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 45 | 41 | 7 | 9
Pain (General disorders) | 0 | 1 | 1 | 2
Pelvic mass (General disorders) | 1 | 0 | 0 | 0
Perforated ulcer (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 25 | 13 | 4 | 3
Spinal pain (General disorders) | 1 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 19 | 13 | 4 | 3
Sudden death (General disorders) | 20 | 16 | 9 | 4
Swelling (General disorders) | 0 | 1 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 2 | 1 | 0 | 0
Ulcer (General disorders) | 1 | 0 | 0 | 0
Ulcer haemorrhage (General disorders) | 1 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 2 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 7 | 3 | 0 | 2
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 3 | 0 | 0 | 1
Biliary cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 6 | 2 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 2 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 13 | 12 | 3 | 6
Cholecystitis acute (Hepatobiliary disorders) | 8 | 11 | 1 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 3 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 13 | 20 | 4 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic artery aneurysm (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 7 | 4 | 0 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 3 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 3 | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0
Contrast media allergy (Immune system disorders) | 2 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 3 | 0 | 0
Iodine allergy (Immune system disorders) | 1 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 1 | 0
Secondary immunodeficiency (Immune system disorders) | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 2 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 2 | 6 | 2 | 0
American trypanosomiasis (Infections and infestations) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 2 | 3 | 1 | 0
Appendiceal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 5 | 2 | 3 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 1 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 2 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 3 | 2 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Biliary abscess (Infections and infestations) | 1 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Bone abscess (Infections and infestations) | 1 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 22 | 22 | 4 | 11
Bronchitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 21 | 22 | 6 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Carbuncle (Infections and infestations) | 2 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 41 | 41 | 16 | 10
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | 0
Chronic hepatitis B (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 3 | 2 | 2 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 2 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis klebsiella (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 10 | 5 | 2 | 1
Device related sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Diabetic foot infection (Infections and infestations) | 5 | 2 | 1 | 0
Diabetic gangrene (Infections and infestations) | 4 | 4 | 0 | 3
Diarrhoea infectious (Infections and infestations) | 2 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 4 | 8 | 2 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0
Emphysematous pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 5 | 2 | 0 | 4
Endocarditis bacterial (Infections and infestations) | 2 | 0 | 0 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 0
Endotoxic shock (Infections and infestations) | 0 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 1 | 0 | 0
Enteritis necroticans (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 18 | 15 | 6 | 6
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 2 | 2 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0
Gallbladder abscess (Infections and infestations) | 2 | 0 | 0 | 0
Gangrene (Infections and infestations) | 14 | 23 | 0 | 2
Gas gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 32 | 23 | 7 | 8
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 2 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 2 | 0 | 0
HIV infection (Infections and infestations) | 0 | 1 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 6 | 6 | 4 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0 | 0
Infected bites (Infections and infestations) | 1 | 0 | 0 | 0
Infected bunion (Infections and infestations) | 0 | 1 | 0 | 0
Infected fistula (Infections and infestations) | 1 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 6 | 8 | 3 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0
Infective spondylitis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 3 | 1 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 1 | 1
Keratitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Listeria sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 4 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 7 | 8 | 3 | 4
Localised infection (Infections and infestations) | 14 | 10 | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 10 | 6 | 5 | 3
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 21 | 22 | 6 | 2
Lymph node tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 1 | 3 | 0 | 0
Mastoid abscess (Infections and infestations) | 1 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Myelitis (Infections and infestations) | 0 | 1 | 0 | 0
Myiasis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 2 | 3 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 2 | 2 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 20 | 17 | 3 | 8
Osteomyelitis chronic (Infections and infestations) | 1 | 3 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 2 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 1 | 0 | 0
Perihepatic abscess (Infections and infestations) | 2 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 6 | 4 | 1 | 3
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 121 | 100 | 42 | 39
Pneumonia bacterial (Infections and infestations) | 2 | 3 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 4 | 1 | 0 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 3 | 7 | 0 | 0
Prostate infection (Infections and infestations) | 1 | 0 | 1 | 1
Proteus infection (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 1 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 4 | 1 | 0 | 0
Purulent discharge (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 10 | 3 | 4 | 3
Pyelonephritis acute (Infections and infestations) | 5 | 8 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 2 | 0 | 1
Pyonephrosis (Infections and infestations) | 1 | 0 | 0 | 0
Q fever (Infections and infestations) | 1 | 0 | 0 | 0
Renal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory moniliasis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 11 | 13 | 2 | 6
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 1 | 0
Schistosomiasis liver (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 28 | 27 | 9 | 18
Septic encephalopathy (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 15 | 14 | 5 | 7
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1
Sinusitis fungal (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 4 | 0 | 1
Soft tissue infection (Infections and infestations) | 3 | 3 | 0 | 0
Splenic abscess (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 5 | 2 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2 | 4 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 4 | 2 | 2 | 2
Syphilis (Infections and infestations) | 1 | 0 | 0 | 0
Tongue abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 2 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 1 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculous pleurisy (Infections and infestations) | 0 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Ureteritis (Infections and infestations) | 0 | 1 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 56 | 44 | 10 | 15
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 5 | 14 | 4 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 2 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 6 | 1 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 3 | 4 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 3 | 2 | 2
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 1 | 3
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 23 | 10 | 2 | 5
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 8 | 9 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 7 | 13 | 4 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 4 | 2 | 0 | 1
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 7 | 6 | 1 | 5
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 9 | 14 | 3 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 10 | 8 | 0 | 2
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 4 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 4 | 1 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 9 | 4 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 9 | 6 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 2 | 1 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 6 | 3 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Suture rupture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 10 | 3 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic shock (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 5 | 5 | 0 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 1 | 0 | 0
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 20 | 15 | 5 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 3 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 3 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram ambulatory abnormal (Investigations) | 0 | 1 | 0 | 0
Glomerular filtration rate abnormal (Investigations) | 1 | 0 | 0 | 0
HIV test positive (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 1 | 0
Occult blood (Investigations) | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 3
Urinary sediment present (Investigations) | 1 | 0 | 0 | 0
Urine output decreased (Investigations) | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 3 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 26 | 16 | 5 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 44 | 49 | 11 | 8
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 39 | 36 | 9 | 10
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 6 | 5 | 5 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 6 | 5 | 4 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2
Gout (Metabolism and nutrition disorders) | 10 | 12 | 3 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 43 | 45 | 8 | 11
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 44 | 22 | 8 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 66 | 57 | 18 | 15
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 7 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 11 | 2 | 5
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0
Insulin resistance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 6 | 5 | 0 | 3
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 5 | 0 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 4 | 2 | 4 | 1
Shock hypoglycaemic (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Sodium retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 8 | 7 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 10 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 1 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone formation increased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Inguinal mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 9 | 11 | 1 | 5
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 7 | 11 | 0 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 24 | 35 | 2 | 2
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 3 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 6 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 3 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8 | 1 | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8 | 5 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 0
Breast adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 2 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 2 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9 | 2 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endocrine neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 8 | 2 | 3
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6 | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 11 | 2 | 3
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 1 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 2
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 19 | 2 | 8
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 3 | 2
Rectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 3 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3 | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Soft tissue cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Splenic neoplasm malignancy unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4 | 0 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 0 | 1
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Apallic syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 2 | 1 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 1 | 0 | 0
Autonomic neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 2 | 0 | 0 | 0
Basilar artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0
Brain hypoxia (Nervous system disorders) | 0 | 0 | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 2 | 1 | 0 | 0
Brain stem haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 2 | 1 | 1 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery disease (Nervous system disorders) | 1 | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 10 | 18 | 3 | 4
Carotid sinus syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 2 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 3 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 11 | 11 | 4 | 2
Cerebral infarction (Nervous system disorders) | 30 | 27 | 4 | 10
Cerebral ischaemia (Nervous system disorders) | 7 | 1 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 93 | 66 | 23 | 22
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 1 | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 2 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 3 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Coma (Nervous system disorders) | 4 | 4 | 0 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1
Complicated migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 5 | 3 | 1 | 2
Dementia (Nervous system disorders) | 2 | 0 | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Demyelination (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0 | 0 | 0
Diabetic autonomic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Diabetic coma (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 2 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 11 | 12 | 2 | 6
Dizziness (Nervous system disorders) | 19 | 12 | 2 | 1
Dysarthria (Nervous system disorders) | 1 | 3 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 1 | 0 | 0
Encephalitis (Nervous system disorders) | 2 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 2 | 1 | 0
Epidural lipomatosis (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 7 | 4 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 2 | 2 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 3 | 5 | 1 | 1
Headache (Nervous system disorders) | 9 | 5 | 1 | 3
Hemianopia homonymous (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 8 | 5 | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 2 | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 2 | 4 | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 3 | 2 | 2 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 2 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 17 | 15 | 3 | 6
Lacunar infarction (Nervous system disorders) | 8 | 6 | 2 | 1
Lateral medullary syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 7 | 3 | 0 | 3
Lumbar radiculopathy (Nervous system disorders) | 2 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 2 | 2 | 2 | 0
Monoparesis (Nervous system disorders) | 0 | 2 | 0 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0
Motor neurone disease (Nervous system disorders) | 0 | 1 | 0 | 0
Movement disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 1 | 0
Myelitis transverse (Nervous system disorders) | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 2 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 3 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 3 | 0 | 1
Neuroglycopenia (Nervous system disorders) | 2 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 1 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 1 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 3 | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 2 | 0 | 0
Parkinsonism (Nervous system disorders) | 2 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 2 | 1 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 5 | 3 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 1 | 1 | 1
Sciatica (Nervous system disorders) | 3 | 7 | 2 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 0
Simple partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal claudication (Nervous system disorders) | 1 | 2 | 0 | 0
Spinal cord haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord oedema (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 5 | 4 | 3 | 0
Subdural effusion (Nervous system disorders) | 1 | 0 | 0 | 0
Subdural hygroma (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 40 | 33 | 7 | 6
Thalamic infarction (Nervous system disorders) | 3 | 1 | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0 | 1 | 0
Thoracic outlet syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 24 | 25 | 4 | 9
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Ulnar neuritis (Nervous system disorders) | 0 | 1 | 0 | 0
Uraemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 4 | 1 | 1 | 1
Vascular encephalopathy (Nervous system disorders) | 1 | 2 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 6 | 1 | 1 | 3
Vocal cord paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1
Anger (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 9 | 3 | 2 | 1
Delirium (Psychiatric disorders) | 3 | 2 | 0 | 0
Depression (Psychiatric disorders) | 3 | 2 | 0 | 3
Disorientation (Psychiatric disorders) | 1 | 1 | 0 | 0
Echopraxia (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 4
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychogenic pain disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 1 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Social avoidant behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Transient psychosis (Psychiatric disorders) | 0 | 2 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 2 | 2 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Anuria (Renal and urinary disorders) | 2 | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 4 | 4 | 2 | 4
Bladder cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 7 | 3 | 2 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Diabetic end stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 60 | 57 | 14 | 14
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 7 | 10 | 2 | 3
Henoch-Schonlein purpura nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 4 | 3 | 1 | 0
Hydroureter (Renal and urinary disorders) | 0 | 1 | 1 | 0
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 6 | 2 | 1 | 1
Nephropathy (Renal and urinary disorders) | 3 | 1 | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 6 | 8 | 2 | 2
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 2 | 4 | 1 | 1
Oliguria (Renal and urinary disorders) | 3 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 2 | 1 | 0
Renal amyloidosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 3 | 0 | 1
Renal colic (Renal and urinary disorders) | 3 | 4 | 0 | 0
Renal cyst (Renal and urinary disorders) | 2 | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 45 | 24 | 11 | 15
Renal failure acute (Renal and urinary disorders) | 73 | 56 | 27 | 23
Renal failure chronic (Renal and urinary disorders) | 74 | 53 | 26 | 33
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal hypertension (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 84 | 64 | 15 | 13
Renal mass (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Ureteral polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 3 | 5 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 2 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 6 | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 5 | 7 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 3 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 13 | 18 | 4 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatic disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 5 | 1 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Urogenital prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 2 | 0 | 0
Vaginal cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulval oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 19 | 17 | 7 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 4 | 3
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 1 | 0
Asthma late onset (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 29 | 23 | 16 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 | 52 | 11 | 10
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 2 | 2
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 5 | 7
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 11 | 5 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 22 | 13 | 4 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 29 | 12 | 10 | 9
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 12 | 10 | 3 | 4
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper airway resistance syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 8 | 5 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Diabetic dermopathy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 23 | 22 | 4 | 7
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 35 | 21 | 5 | 3
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Activities of daily living impaired (Social circumstances) | 1 | 0 | 0 | 0
Drug abuser (Social circumstances) | 0 | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 3 | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 8 | 5 | 1 | 1
Aortic aneurysm rupture (Vascular disorders) | 2 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0
Aortic rupture (Vascular disorders) | 0 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 5 | 4 | 2 | 2
Arterial disorder (Vascular disorders) | 4 | 2 | 0 | 0
Arterial insufficiency (Vascular disorders) | 0 | 1 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 2 | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 2 | 1 | 0
Arteriosclerosis (Vascular disorders) | 4 | 7 | 0 | 1
Arteriosclerosis Moenckeberg-type (Vascular disorders) | 1 | 0 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0 | 0 | 0
Blood pressure inadequately controlled (Vascular disorders) | 4 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 6 | 5 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 8 | 5 | 5 | 0
Diabetic macroangiopathy (Vascular disorders) | 0 | 0 | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 1 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 1 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 2 | 0 | 2
Femoral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Femoral artery embolism (Vascular disorders) | 0 | 2 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 3 | 1 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 6 | 2 | 2 | 1
Haemodynamic instability (Vascular disorders) | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 38 | 47 | 7 | 13
Hypertensive crisis (Vascular disorders) | 14 | 18 | 3 | 3
Hypertensive emergency (Vascular disorders) | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 31 | 32 | 3 | 11
Hypovolaemic shock (Vascular disorders) | 3 | 2 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 1 | 0 | 0
Infarction (Vascular disorders) | 1 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 10 | 8 | 1 | 2
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Labile hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Leriche syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 2 | 1 | 0 | 0
Neovascularisation (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 12 | 8 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 23 | 31 | 8 | 10
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 9 | 13 | 3 | 4
Peripheral circulatory failure (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 2 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 13 | 11 | 2 | 2
Peripheral vascular disorder (Vascular disorders) | 5 | 10 | 1 | 3
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 3 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian steal syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 1 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Varicophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Varicose ulceration (Vascular disorders) | 1 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 2 | 0 | 1
Vascular stenosis (Vascular disorders) | 1 | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 1 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 2 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core-phase: Aliskiren (N=4272) | Core-phase: Placebo (N=4285) | Extension-phase: Aliskiren (N=3773) | Extension-phase: Placebo (N=3817)
Anaemia (Blood and lymphatic system disorders) | 270 | 270 | 94 | 76
Constipation (Gastrointestinal disorders) | 202 | 241 | 48 | 45
Diarrhoea (Gastrointestinal disorders) | 405 | 305 | 56 | 41
Oedema peripheral (General disorders) | 655 | 670 | 130 | 112
Bronchitis (Infections and infestations) | 217 | 211 | 36 | 61
Nasopharyngitis (Infections and infestations) | 398 | 369 | 83 | 89
Upper respiratory tract infection (Infections and infestations) | 214 | 215 | 48 | 58
Urinary tract infection (Infections and infestations) | 286 | 243 | 72 | 88
Hyperkalaemia (Metabolism and nutrition disorders) | 1650 | 1229 | 270 | 252
Hypoglycaemia (Metabolism and nutrition disorders) | 334 | 297 | 98 | 87
Arthralgia (Musculoskeletal and connective tissue disorders) | 295 | 299 | 52 | 51
Back pain (Musculoskeletal and connective tissue disorders) | 360 | 344 | 54 | 46
Pain in extremity (Musculoskeletal and connective tissue disorders) | 292 | 311 | 57 | 42
Dizziness (Nervous system disorders) | 314 | 305 | 45 | 57
Headache (Nervous system disorders) | 188 | 219 | 42 | 28
Renal impairment (Renal and urinary disorders) | 352 | 321 | 72 | 87
Cough (Respiratory, thoracic and mediastinal disorders) | 256 | 280 | 53 | 47
Hypertension (Vascular disorders) | 380 | 410 | 121 | 105
Hypotension (Vascular disorders) | 496 | 321 | 34 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.